CLINICAL TRIAL: NCT07308782
Title: An Exploratory Pharmacodynamic Clinical Study of CL-197 Capsules in Treatment Naive Patients With Human Immunodeficiency Virus (HIV-1)
Brief Title: A Phase Ⅱa Clinical Study of CL-197 Capsules
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Genuine Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GB-CL-197-102
Record Dates: First submitted 2025-11-26; First posted 2025-12-30 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: HIV-1 Infection
Keywords: HIV-1 infection; CL-197

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CL-197 capsules (Experimental)
  Interventions: Drug: CL-197 capsules

INTERVENTIONS:
Drug: CL-197 capsules — Participants will take a single dose of CL-197 capsules at a dose of 10 mg, 30 mg or 60 mg, orally on an empty stomach.

SUMMARY:
This study will evaluate the antiretroviral activity, safety and pharmacokinetics of single dose of CL-197 capsule in three dose groups administered to antiretroviral treatment-naïve adult participants with human immunodeficiency virus type 1 (HIV-1) infection.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 18-60 (including boundary values), both male and female.
2. Body mass index (BMI) range between 18.5-29.9 (including the boundary value). Body weight ≥ 50.0 kg for men and ≥ 45.0 kg for women.
3. Participants diagnosed with HIV-1 infection before screening, and never received any anti-HIV drugs or HIV-related vaccine therapy (including investigational or other unmarketed anti-HIV drugs or vaccines) before screening.
4. Participants who agree not to receive other anti-HIV drugs during the trial period (from signing the informed consent form until the Day 13 sampling).
5. CD4 cell count > 200 cells/μL at screening.
6. Women of childbearing potential (WOCBP) must have adopted effective non-drug contraceptive measures, have a negative serum pregnancy test at screening/baseline, and be willing to use appropriate effective methods of contraception from signing the informed consent form until 3 months after the last dose of the study drug. Male study participants must be willing to refrain from fathering children and voluntarily use effective contraception during the trial and until 3 months after the last dose of the study drug, or have been surgically sterilized.
7. Participants who understand and sign the informed consent form.

Exclusion Criteria:

1. Diagnosis of acute HIV-1 infection, or presence of an AIDS-defining disease at enrollment, or history of an opportunistic infection within 3 months prior to enrollment with the condition remaining unstable within 4 weeks prior to enrollment.
2. Had pre-exposure prophylaxis (PrEP) and/or post-exposure prophylaxis (PEP) treatment within 1 month prior to screening.
3. Had any clinically significant disease (including cardiovascular, respiratory, digestive, endocrine/metabolic, neurological/psychiatric, hematological, and immune system diseases, etc.) that is poorly controlled, as determined by the investigator at screening.
4. Resting systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg, or heart rate > 100 beats per minute, or heart rate < 50 beats per minute, or QTcF (QT interval corrected for heart rate according to Fridericia's formula) > 450 ms, or fasting blood glucose ≥ 7.0 mmol/L.
5. History of severe allergy (immediate, life-threatening systemic anaphylaxis) to drugs (e.g., aspirin or cephalosporin antibiotics), other drug components (e.g., lactose or gelatin), or food, or history of allergic diseases requiring medication control (e.g., asthma, urticaria, atopic dermatitis/eczema, etc.) prior to screening.
6. Had major gastrointestinal surgery within 6 months prior to screening (except uncomplicated appendectomy or cholecystectomy), or any surgery that could affect drug absorption, distribution, metabolism and excretion; or planned elective surgery during the trial period, as determined by the investigator at screening.
7. History of malignancy (except carcinoma in situ of the cervix treated with conization, or radically resected basal cell carcinoma, squamous cell carcinoma, and/or carcinoma in situ [Bowen's disease] of the skin).
8. Hepatitis B surface antigen (HBsAg) positive at screening, or active syphilis, or Hepatitis C virus (HCV) antibody positive, or previous interferon treatment for HBV infection leading to HBsAg seroconversion.
9. Hemoglobin (Hb) < 110 g/L, or white blood cell (WBC) count < 3 × 10^9/L, or absolute neutrophil count (ANC) < 1 × 10^9/L, or platelet (PLT) count < 100 × 10^9/L at screening.
10. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≥ 2.5 times upper limit of normal (ULN), or total bilirubin (TBIL) ≥ 1.5 × ULN at screening.
11. Serum creatinine (SCr) > 1.1 × ULN, or creatinine clearance (Ccr) < 60 mL/min (calculated by Cockcroft-Gault formula) at screening.
12. Participants smoke more than 5 cigarettes daily on average within 3 months prior to screening, or may be unwilling to stop using any tobacco products during drug administration and sampling periods.
13. Drinking more than 14 units of alcohol (1 unit of alcohol ≈ 360 mL of beer with 5% alcohol, or 45 mL of liquor with 40% alcohol, or 150 mL of wine with 12% alcohol) within 3 months prior to screening on average, or positive alcohol breath test at screening or baseline, or unwillingness to stop using any alcohol-containing products during hospitalization.
14. Excessive consumption of tea, coffee, and/or caffeine-containing beverages (averaging more than 8 cups per day, 1 cup ≈ 250 mL) within 3 months prior to screening on average, or unwillingness to stop consuming tea, coffee, and/or caffeine-containing beverages during hospitalization.
15. Participants with consumption of pitaya, mango, pomelo, carambola, or foods/beverages prepared from them, or foods/beverages containing xanthine, caffeine, or alcohol (including chocolate, tea, coffee, cola, cocoa, etc.), or any other special diet that may affect drug absorption, distribution, metabolism, or excretion within 48 hours prior to the first dose of the investigational product, or unwillingness to stop using them during hospitalization.
16. History of drug abuse (non-medical, excessive, misuse, or addictive use of any drug leading to social, psychological, or physical impairment) within 5 years prior to screening, or positive urine drug screen at screening or baseline.
17. Intolerance to venipuncture, or history of needle or blood phobia, or blood donation (including component blood) or significant blood loss (≥400 mL) or blood transfusion within 3 months prior to screening, or blood donation plan during the trial.
18. Specific dietary requirements during the trial, or inability to accept the standardized diet.
19. Have participated in or are participating in other investigational drug or interventional medical device clinical trials (having signed informed consent and received investigational drug/interventional device or placebo) within 3 months prior to screening.
20. Pregnant or breastfeeding females at screening, or positive serum pregnancy test (applicable to WOCBP only).
21. Have a birth plan (including egg or sperm donation) by WOCBP or male participants from 1 month prior to informed consent until 3 months after administration of the investigational drug, or unwillingness to use effective contraception/barrier methods (including one or more non-drug contraceptive methods or abstinence from heterosexual activity).
22. Use of any prescription drugs, over-the-counter drugs, Chinese herbal medicines, or health products within 14 days prior to dosing.
23. Any other conditions considered by the investigator as unsuitable for participation in this trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-11-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in log10 value of HIV-1 Ribonucleic acid (RNA) on Day 8 | Baseline and Day 8.

SECONDARY OUTCOMES:
Change from baseline in log10 value of HIV-1 RNA on Day 11 | Baseline and Day 11.
Change from baseline in CD4+ cell count on Day 13 | Baseline and Day 13.
Incidence of adverse events (AEs) / serious AEs | Day 13.
  AEs are assessed based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table).
Time to Maximum Concentration (Tmax) of CL -197 | Up to 13 days post-dose.
Elimination Half-Life (t1/2) of CL -197 | Up to 13 days post-dose.
Maximum Observed Plasma Concentration (Cmax) of CL -197 | Up to 13 days post-dose.
Area Under the Concentration-time Curve (AUC) of CL -197 | Up to 13 days post-dose.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Youan Hospital, Capital Medical University, Beijing, China